CLINICAL TRIAL: NCT04148144
Title: Low Back Pain Among Care-seeking Families in General Practice (The YoungBack Project): a Prospective Parallel Cohort Study in 400 Children and Adolescents and Their Parents
Brief Title: Low Back Pain Among Care-seeking Families in General Practice
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: University College of Northern Denmark (Other)
Responsible Party: Principal Investigator, Christian Lund Straszek, Principal Investigator, Aalborg University
Other Study IDs: The YoungBack Project
Record Dates: First submitted 2019-10-24; First posted 2019-11-01 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Low Back Pain
Keywords: Low back pain; Adolescent; Parent; Prognosis; General practice
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents with low back pain: Adolescents aged 8-19 with low back pain.
  Interventions: Other: No intervention included
- Parents of included adolescents: Parents recruited for the parallel cohort, are required to be a parent or a legal guardian of the included adolescent. Siblings, grandparents or a similar person are not eligible for inclusion in the parallel cohort.
  Interventions: Other: No intervention included

INTERVENTIONS:
Other: No intervention included — No intervention included

SUMMARY:
Background Low back pain (LBP) is the largest cause of years lived with disability worldwide and often associated with low quality of life, inability to work and low physical activity levels. In Danish general practice, LBP accounts for nearly 10% of all yearly consultations, making it the number one reason for consulting a general practitioner in Denmark. An increase in care-seeking children and adolescents with LBP in general practice is seen in the pre-teen-age-years.

At present, no study has investigated on the natural prognosis of LBP among care-seeking adolescents in general practice. Furthermore, the potential impact of patient and parent-related factors on prognosis remains unknown. The aims of the study are to 1) investigate the natural prognosis of LBP and 2) identify patient and parent-related factors which my influence prognosis.

Methods Adolescents aged 8 to 19 years consulting their general practitioner due to LBP will be invited to participate in this prospective cohort study. One parent of each patient will be invited to be a part of the parallel cohort. Online questionnaires will be used to collect data on patient characterises, pain intensity, pain frequency, medication, health-related quality of life, physical activity and illness perception at baseline and at the one-year follow-up. Data on pain intensity and parent-related worries will be collected through biweekly text messages. LBP will be assessed by latent class analysis.

Discussion This study will be the first to uncover the natural prognosis of LBP within a young, care-seeking population in general practice and to investigate if factors related to the patient or parents influence prognosis.

ELIGIBILITY:
Inclusion Criteria:

For adolescents in the primary cohort:

* age between 8 and 19
* experiencing low back pain

For parents in the parallel cohort:

- parent or legal guardian of included adolescents

Exclusion Criteria:

- not providing informed consent.

Ages: 8 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents with low back pain in Danish general practice and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Worst low back pain during the week prior to consulting the general practitioner. | At 12 month
  Is measured on an 100mm visual analogue scale (0mm equals no pain and 100mm equals worst possible pain).
  Only the adolescents with LBP from the primary cohort is asked this question.

SECONDARY OUTCOMES:
LBP frequency | At baseline and after 12 month
  Response: 5-point Likert scale (daily, several times per week, weekly, monthly, rarely).
  Only the adolescents with LBP from the primary cohort is asked this question.
LBP affecting participation in usual daily activities | At baseline and every month for 12 month
  Response: yes/no. Only the adolescents with LBP from the primary cohort is asked this question.
Health-related quality of life - psychologic wellbeing | At baseline and after 12 month
  Question: "Have you felt satisfied with your life?" Response: not at all, slightly, moderately, very and extremely Only the adolescents with LBP from the primary cohort is asked this question.
Health-related quality of life - moods and emotions | At baseline and after 12 month
  Question: Have you felt under pressure? Response: never, seldom, quite often, very often, always Only the adolescents with LBP from the primary cohort is asked this question.
Illness perception (adolescent) | At baseline and every month for 12 month
  Question: Are you worried about your back pain? Response: 10-point scale with 0 being equal to "not worried at all" whereas 10 will be equal to "very worried".
  Only the adolescents with LBP from the primary cohort is asked this question.
Sleep | At baseline and every month for 12 month
  Question: How many hours do you sleep on average during the night? Response: hours/night Both adolescents and parents are asked this question.
Pain interference | At baseline and every month for 12 month
  Response: I have no problems doing my usual activities, I have slight problems doing my usual activities, I have moderate problems doing my usual activities, I have severe problems doing my usual activities or I have extreme problems doing my usual activities.
  Only the adolescents with LBP from the primary cohort is asked this question.
LBP within the week prior to being enrolled in the study | At baseline
  Response: yes/no
  Only parents from the parallel cohort is asked this question.
Health-related quality of life (parent) | At baseline
  Euroqol 5 dimensions 5 levels (EQ-5D-5L) questionnaire
  Only parents from the parallel cohort is asked these question.
Illness perception (parent) | At baseline
  Question: Are you worried about your child's back pain? Response: 10-point scale with 0 being equal to "not worried at all" whereas 10 will be equal to "very worried".
  Only parents from the parallel cohort is asked this question.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for General Practice at Aalborg University, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided